CLINICAL TRIAL: NCT02162667
Title: Phase 3 Efficacy and Safety Study of CT-P6 and Herceptin as Neoadjuvant and Adjuvant Treatment in Patients With Her2-positive Early Breast Cancer
Brief Title: Efficacy and Safety Evaluating Study of CT-P6 in Her2 Positive Early Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celltrion (Industry)
Collaborators: Nippon Kayaku Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CT-P6 3.2; 2013-004525-84 (EudraCT Number)
Record Dates: First submitted 2014-06-11; First posted 2014-06-13 (Estimated); Results first posted 2019-10-29 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2019-10

CONDITIONS: HER2-positive Carcinoma of Breast
MeSH Terms: interventions — Trastuzumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CT-P6 (Experimental)
  Interventions: Drug: Trastuzumab
- Trastuzumab (Active Comparator)
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: Trastuzumab — Trastuzumab 6mg/kg is ongoing to be administered for both arms after 8mg/kg loading dose.
  Other Names: Herceptin

SUMMARY:
This study will determine whether CT-P6 and Herceptin are equivalent in patients with early-stage breast cancer undergoing neoadjuvant chemotherapy. Our hypothesis is that the pathologic complete response rate will be equivalent in patients treated with neoadjuvant CT-P6 or Herceptin. Patients will receive 8 cycles of neoadjuvant systemic therapy and up to 10 cycles of therapy in the adjuvant setting.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has histologically confirmed and newly diagnosed breast cancer
* Patient who has clinical stage I, II, or IIIa operable breast cancer according to AJCC (American Joint Committee on Cancer) Breast Cancer Staging 7th edition
* Patient who has HER2-positive status confirmed locally, defined as 3+ score by IHC (immuno-histochemistry).

Exclusion Criteria:

* Patient who has bilateral breast cancer
* Patient who has received prior treatment for breast cancer, including chemotherapy, biologic therapy, hormone therapy, immunotherapy, radiation or surgery, including any prior therapy with anthracyclines.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 562 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-05-26 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (83):
- Argentina (6):
  - Buenos Aires
  - Córdoba
  - Quilmes
  - Rosario
  - San Salvador de Jujuy
  - Santa Rosa
- Belarus (2):
  - Brest
  - Minsk
- Sarajevo, Bosnia and Herzegovina
- Chile (2):
  - Santiago
  - Temuco
- Nancy, France
- Tbilisi, Georgia
- Hungary (2):
  - Budapest
  - Debrecen
- India (9):
  - Bangalore
  - Chennai
  - Delhi
  - Jaipur
  - Kolkata
  - Mumbai
  - Nashik
  - New Delhi
  - Pune
- Italy (4):
  - Bari
  - Pavia
  - Piacenza
  - Rimini
- Tokyo, Japan
- Latvia (2):
  - Daugavpils
  - Riga
- Mexico (2):
  - Acapulco
  - Monterrey
- Peru (3):
  - Arequipa
  - Lima
  - Trujillo
- Philippines (7):
  - Cebu
  - City of Taguig
  - Makati
  - Manila
  - Pasig
  - Quezon City
  - San Juan City
- Poland (3):
  - Gdansk
  - Lodz
  - Warsaw
- Lisbon, Portugal
- Romania (4):
  - Brasov
  - Bucharest
  - Cluj-Napoca
  - Suceava
- Russia (12):
  - Arkhangelsk
  - Kazan'
  - Krasnoyarsk
  - Kursk
  - Moscow
  - Nizhny Novgorod
  - Novosibirsk
  - Obninsk
  - Omsk
  - Saint Petersburg
  - Samara
  - Saransk
- South Africa (5):
  - Cape Town
  - George
  - Johannesburg
  - Port Elizabeth
  - Pretoria
- Spain (2):
  - Seville
  - Zaragoza
- Taiwan (3):
  - Kaohsiung City
  - Taichung
  - Taipei
- Ukraine (10):
  - Cherkasy
  - Donetsk
  - Kharkiv
  - Kherson
  - Khmelnytskyi
  - Poltava
  - Sumy
  - Uzhhorod
  - Vinnytsia
  - Zaporizhzhia

REFERENCES:
- [Derived] Stebbing J, Baranau YV, Baryash V, Manikhas A, Moiseyenko V, Dzagnidze G, Zhavrid E, Boliukh D, Pikiel J, Eniu AE, Li RK, Tiangco B, Lee SJ, Kim S. Long-term efficacy and safety of CT-P6 versus trastuzumab in patients with HER2-positive early breast cancer: final results from a randomized phase III trial. Breast Cancer Res Treat. 2021 Aug;188(3):631-640. doi: 10.1007/s10549-021-06240-5. Epub 2021 Jun 20. PMID 34148205
- [Derived] Esteva FJ, Baranau YV, Baryash V, Manikhas A, Moiseyenko V, Dzagnidze G, Zhavrid E, Boliukh D, Stroyakovskiy D, Pikiel J, Eniu AE, Li RK, Rusyn AV, Tiangco B, Lee SJ, Lee SY, Yu SY, Stebbing J. Efficacy and safety of CT-P6 versus reference trastuzumab in HER2-positive early breast cancer: updated results of a randomised phase 3 trial. Cancer Chemother Pharmacol. 2019 Oct;84(4):839-847. doi: 10.1007/s00280-019-03920-4. Epub 2019 Aug 19. PMID 31428820
- [Derived] Stebbing J, Baranau Y, Baryash V, Manikhas A, Moiseyenko V, Dzagnidze G, Zhavrid E, Boliukh D, Stroyakovskii D, Pikiel J, Eniu A, Komov D, Morar-Bolba G, Li RK, Rusyn A, Lee SJ, Lee SY, Esteva FJ. CT-P6 compared with reference trastuzumab for HER2-positive breast cancer: a randomised, double-blind, active-controlled, phase 3 equivalence trial. Lancet Oncol. 2017 Jul;18(7):917-928. doi: 10.1016/S1470-2045(17)30434-5. Epub 2017 Jun 4. PMID 28592386

RESULTS

PARTICIPANT FLOW:
Groups:
- CT-P6: Patient received CT-P6 at an initial dose of 8 mg/kg administered by a single IV infusion on Day 1 of Cycle 1, followed by 6 mg/kg on Day 1 of Cycles 2 through 8 (3-week cycles). Patients also received docetaxel 75 mg/m^2 during cycles 1 through 4 and FEC (fluorouracil 500mg/m^2, epirubicin 75mg/m^2, and cyclophosphamide 500mg/m^2) during Cycles 5 through 8. After a total of 8 treatment cycles of the neoadjuvant treatment, surgery was performed within 3 to 6 weeks from the last dose of study in the neoadjuvant period. Three to 6 weeks after surgery, patients entered the adjuvant period and received additional CT-P6 6 mg/kg (3-week cycles) for up to 1 year from the first day of study drug administration in the Neoadjuvant Period, excluding surgery (or up to 10 cycles after surgery)
- Herceptin: Patient received Herceptin at an initial dose of 8 mg/kg administered by a single IV infusion on Day 1 of Cycle 1, followed by 6 mg/kg on Day 1 of Cycles 2 through 8 (3-week cycles). Patients also received docetaxel 75 mg/m^2 during cycles 1 through 4 and FEC (fluorouracil 500mg/m^2, epirubicin 75mg/m^2, and cyclophosphamide 500mg/m^2) during Cycles 5 through 8. After a total of 8 treatment cycles of the neoadjuvant treatment, surgery was performed within 3 to 6 weeks from the last dose of study in the neoadjuvant period. Three to 6 weeks after surgery, patients entered the adjuvant period and received additional Herceptin 6 mg/kg (3-week cycles) for up to 1 year from the first day of study drug administration in the Neoadjuvant Period, excluding surgery (or up to 10 cycles after surgery).
Period: Neoadjuvant Period
Arm/Group | CT-P6 | Herceptin
Started | 278 | 284
Completed (the number of patients who completed 8 cycles of the Neoadjuvant Period and underwent surgery.) | 264 | 267
Not Completed | 14 | 17
Period: Adjuvant Period
Arm/Group | CT-P6 | Herceptin
Started | 260 | 268
Completed | 248 | 255
Not Completed | 12 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CT-P6 | Herceptin | Total
Number analyzed (Participants) | 278 | 284 | 562
Age, Continuous [Median (Full Range); unit: years] | 53.0 [24 to 79] | 52.5 [22 to 74] | 53.0 [22 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 278 | 284 | 562
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients Achieving Pathological Complete Response Defined as the Absence of Invasion Tumor Cells in the Breast and in Axillary Lymph Nodes, Regardless of Ductal Carcinoma in Situ (DCIS)
Description: Subject who went through Neoadjuvant period completely (24 weeks), will receive surgery within 3-6 weeks after last treatment of neoadjuvant period.
  The primary endpoint, Pathological complete response, will be assessed using resected bio-specimens collected in breast and axilla during a surgery.
Time Frame: After Neo-adjuvant therapy and Surgery (up to 30 weeks)
Population: Per-Protocol Set: All patients randomly assigned to study drug, regardless of whether or not any study treatment dosing is completed, except for those patients excluded because of major protocol deviations.
Measure: Number (95% Confidence Interval); unit: percentage of responders
Groups:
- CT-P6: Patient received CT-P6 at an initial dose of 8 mg/kg administered by a single IV infusion on Day 1 of Cycle 1, followed by 6 mg/kg on Day 1 of Cycles 2 through 8 (3-week cycles). Patients also received docetaxel 75 mg/m^2 during cycles 1 through 4 and FEC (fluorouracil 500mg/m^2, epirubicin 75mg/m^2, and cyclophosphamide 500mg/m^2) during Cycles 5 through 8. After a total of 8 treatment cycles of the neoadjuvant treatment, surgery was performed within 3 to 6 weeks from the last dose of study.
- Herceptin: Patient received Herceptin at an initial dose of 8 mg/kg administered by a single IV infusion on Day 1 of Cycle 1, followed by 6 mg/kg on Day 1 of Cycles 2 through 8 (3-week cycles). Patients also received docetaxel 75 mg/m^2 during cycles 1 through 4 and FEC (fluorouracil 500mg/m^2, epirubicin 75mg/m^2, and cyclophosphamide 500mg/m^2) during Cycles 5 through 8. After a total of 8 treatment cycles of the neoadjuvant treatment, surgery was performed within 3 to 6 weeks from the last dose of study.
Arm/Group | CT-P6 | Herceptin
Number analyzed (Participants) | 248 | 256
percentage of responders | 46.77 [40.43 to 53.19] | 50.39 [44.10 to 56.68]

2. Secondary Outcome: The Percentage of Patients Achieving Pathological Complete Response (pCR) of the Breast Regardless of DCIS With Positive or Unknown Nodal Status
Description: Subject who went through Neoadjuvant period completely (24 weeks), will receive surgery within 3-6 weeks after last treatment of neoadjuvant period.
  The secondary endpoint, other than pCR of breast and axillary nodes ragardless of DCIS which was primary endpoint, will be assessed using resected bio-specimens collected in breast and axilla during a surgery.
Time Frame: After Neo-adjuvant therapy and Surgery (up to 30 weeks)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | CT-P6 | Herceptin
Number analyzed (Participants) | 248 | 256
percentage of responders | 4.84 [2.52 to 8.30] | 4.69 [2.45 to 8.04]

3. Secondary Outcome: The Percentage of Patients Achieving Pathological Complete Response of the Breast and Axillary Nodes With Absence of DCIS
Description: as for outcome 2
Time Frame: After Neo-adjuvant therapy and Surgery (up to 30 weeks)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | CT-P6 | Herceptin
Number analyzed (Participants) | 248 | 256
percentage of responders | 39.92 [33.78 to 46.31] | 41.41 [35.31 to 47.71]

4. Secondary Outcome: Overall Response Rate (ORR) From Local Review
Description: The ORR was defined as the proportion of patients with a BOR of CR or PR as assessed by RECIST guideline Version 1.1 during the Nedadjuvant Period.
Time Frame: After Neo-adjuvant therapy (up to 24 weeks)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of responders
Groups:
- CT-P6: Patient received CT-P6 at an initial dose of 8 mg/kg administered by a single IV infusion on Day 1 of Cycle 1, followed by 6 mg/kg on Day 1 of Cycles 2 through 8 (3-week cycles). Patients also received docetaxel 75 mg/m^2 during cycles 1 through 4 and FEC (fluorouracil 500mg/m^2, epirubicin 75mg/m^2, and cyclophosphamide 500mg/m^2) during Cycles 5 through 8.
- Herceptin: Patient received Herceptin at an initial dose of 8 mg/kg administered by a single IV infusion on Day 1 of Cycle 1, followed by 6 mg/kg on Day 1 of Cycles 2 through 8 (3-week cycles). Patients also received docetaxel 75 mg/m^2 during cycles 1 through 4 and FEC (fluorouracil 500mg/m^2, epirubicin 75mg/m^2, and cyclophosphamide 500mg/m^2) during Cycles 5 through 8.
Arm/Group | CT-P6 | Herceptin
Number analyzed (Participants) | 248 | 256
percentage of responders | 84.27 [79.14 to 88.57] | 83.98 [78.91 to 88.26]

5. Secondary Outcome: Disease-free Survival
Description: Patients who underwent breast surgery were included in the DFS analysis. Disease-free survival was defined as the interval between the date of breast surgery and disease progression, recurrence, or death from any cause, whichever occurred first. Only a recurrence or progression of disease that occurred before beginning another anticancer therapy was regarded as an event.
Time Frame: Up to 3 years from the day of last patient enrollment (during whole study period)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- CT-P6: Patient received CT-P6 at an initial dose of 8 mg/kg administered by a single IV infusion on Day 1 of Cycle 1, followed by 6 mg/kg on Day 1 of Cycles 2 through 8 (3-week cycles). Patients also received docetaxel 75 mg/m^2 during cycles 1 through 4 and FEC (fluorouracil 500mg/m^2, epirubicin 75mg/m^2, and cyclophosphamide 500mg/m^2) during Cycles 5 through 8. After a total of 8 treatment cycles of the neoadjuvant treatment, surgery was performed within 3 to 6 weeks from the last dose of study. Three to 6 weeks after surgery, patients entered the adjuvant period and received additional CT-P6 6 mg/kg (3-week cycles) for up to 1 year from the first day of study drug administration in the Neoadjuvant Period, excluding surgery (or up to 10 cycles after surgery)
- Herceptin: Patient received Herceptin at an initial dose of 8 mg/kg administered by a single IV infusion on Day 1 of Cycle 1, followed by 6 mg/kg on Day 1 of Cycles 2 through 8 (3-week cycles). Patients also received docetaxel 75 mg/m^2 during cycles 1 through 4 and FEC (fluorouracil 500mg/m^2, epirubicin 75mg/m^2, and cyclophosphamide 500mg/m^2) during Cycles 5 through 8. After a total of 8 treatment cycles of the neoadjuvant treatment, surgery was performed within 3 to 6 weeks from the last dose of study. Three to 6 weeks after surgery, patients entered the adjuvant period and received additional Herceptin 6 mg/kg (3-week cycles) for up to 1 year from the first day of study drug administration in the Neoadjuvant Period, excluding surgery (or up to 10 cycles after surgery).
Arm/Group | CT-P6 | Herceptin
Number analyzed (Participants) | 248 | 256
proportion of participants
  1 year | 0.95 [0.91 to 0.97] | 0.96 [0.93 to 0.98]
  2 years | 0.87 [0.81 to 0.90] | 0.89 [0.85 to 0.92]
  3 years | 0.82 [0.77 to 0.87] | 0.82 [0.75 to 0.88]

6. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival was defined as the interval between randomization and disease progression, recurrence, or death from any cause, whichever occurred first. Only a recurrence or progression of disease that occurred before beginning another anticancer therapy was regarded as an event.
Time Frame: Up to 3 years from the day of last patient enrollment (during whole study period)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | CT-P6 | Herceptin
Number analyzed (Participants) | 248 | 256
proportion of participants
  1 year | 0.99 [0.97 to 1.00] | 0.98 [0.95 to 0.99]
  2 years | 0.90 [0.86 to 0.94] | 0.93 [0.89 to 0.95]
  3 years | 0.82 [0.77 to 0.87] | 0.87 [0.82 to 0.90]

7. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the interval between randomization and death from any cause.
Time Frame: Up to 3 years from the day of last patient enrollment (during whole study period)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | CT-P6 | Herceptin
Number analyzed (Participants) | 248 | 256
proportion of participants
  1 year | 1.00 [1.00 to 1.00] | 1.00 [0.97 to 1.00]
  2 years | 0.98 [0.95 to 0.99] | 0.98 [0.96 to 0.99]
  3 years | 0.95 [0.91 to 0.97] | 0.94 [0.90 to 0.96]

8. Secondary Outcome: The Number of Patients Who Had Progressive Disease or Recurrence
Description: If recurrence or progression of disease occurred at any time during the study, the progressed tumor site was recorded in the "recurrence or progression of disease" eCRF page as local, regional, or distant, with diagnostic method and whether positive cytology or histology or not.
  The resulting recurrence or progression of disease information was summarized as secondary endpoint.
Time Frame: Up to 3 years from the day of last patient enrollment (during whole study period)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | CT-P6 | Herceptin
Number analyzed (Participants) | 248 | 256
participants
  Overall Period | 41 | 35
  Neoadjuvant Period | 1 | 2
  Adjuvant Period | 5 | 3
  Follow-up Period | 35 | 30

9. Secondary Outcome: Maximum Serum Concentration After Administration (Cmax) in Each Cycle
Description: Pharmacokinetic samples were collected before study drug (CT-P6 or US-licensed Herceptin) administration (within 15 minutes prior to the beginning of the study drug infusion) and within 15 minutes after the end of the study drug infusion for each cycle during the Neoadjuvant Period. After the completion of treatment, an additional PK sample was collected at the EOT1.
Time Frame: End of each treatment cycles, up to 24 weeks (during neoadjuvant period)
Population: Safety Analysis Set: All patients randomly assigned to study drug and who receive at least 1 dose (fully or partially) of study drug
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | CT-P6 | Herceptin
Number analyzed (Participants) | 271 | 278
µg/mL
  Cycle 1 | 186.428 (69.0828) | 178.567 (55.3800)
  Cycle 2 | 145.078 (47.7899) | 138.989 (45.7103)
  Cycle 3 | 145.183 (44.5392) | 141.130 (43.8189)
  Cycle 4 | 148.541 (54.2737) | 137.465 (45.6914)
  Cycle 5 | 136.210 (44.6078) | 135.307 (47.1950)
  Cycle 6 | 143.569 (42.4510) | 143.605 (51.2868)
  Cycle 7 | 146.726 (48.0249) | 141.468 (43.1823)
  Cycle 8 | 145.081 (41.5382) | 144.238 (57.3618)

10. Secondary Outcome: Trough Serum Concentration (Ctrough) in Each Cycle
Description: as for outcome 9
Time Frame: Pre-infusion of cycles 1 to 8 during neoadjuvant period
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | CT-P6 | Herceptin
Number analyzed (Participants) | 271 | 278
µg/mL
  Cycle 1 | 18.915 (22.9964) | 18.905 (21.2967)
  Cycle 2 | 17.346 (17.9771) | 16.773 (16.8134)
  Cycle 3 | 16.796 (17.2409) | 17.816 (23.3438)
  Cycle 4 | 17.851 (20.1572) | 15.904 (15.8754)
  Cycle 5 | 18.403 (19.9042) | 17.962 (17.9429)
  Cycle 6 | 18.902 (20.2198) | 18.256 (17.6964)
  Cycle 7 | 18.540 (14.3313) | 18.718 (18.5976)
  Cycle 8 | 17.901 (7.2203) | 17.129 (10.0491)

11. Post Hoc Outcome: The Percentage of Patients Achieving Pathological Complete Response of the Breast and Axillary Nodes Regardless of DCIS
Description: as for outcome 2
Time Frame: After Neo-adjuvant therapy and Surgery (up to 30 weeks)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | CT-P6 | Herceptin
Number analyzed (Participants) | 248 | 256
percentage of responders | 51.61 [45.20 to 57.98] | 55.08 [48.76 to 61.28]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the date the informed consent form is signed until up to 30 days from last dose of study drug, regardless of the relationship to the study drug
Arm/Group | CT-P6 | Herceptin
Serious Adverse Events (participants affected / at risk) | 22/271 | 36/278
Other Adverse Events (participants affected / at risk) | 263/271 | 264/278
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CT-P6 (N=271) | Herceptin (N=278)
Anemia (Blood and lymphatic system disorders) | 1 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 3
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 3
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Adams-Stokes syndrome (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Dacryostenosis acquired (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Implant site extravasation (General disorders) | 1 | 0
Incarcerated hernia (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 2
Endocarditis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 1
Postoperative abscess (Infections and infestations) | 1 | 0
Septic embolus (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Complications of transplant surgery (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1
Scar (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Heart rate irregular (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Oocyte harvest (Surgical and medical procedures) | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CT-P6 (N=271) | Herceptin (N=278)
Anaemia (Blood and lymphatic system disorders) | 59 | 67
Febrile neutropenia (Blood and lymphatic system disorders) | 11 | 16
Leukopenia (Blood and lymphatic system disorders) | 28 | 41
Neutropenia (Blood and lymphatic system disorders) | 95 | 116
Lacrimation increased (Eye disorders) | 16 | 15
Constipation (Gastrointestinal disorders) | 24 | 18
Diarrhoea (Gastrointestinal disorders) | 52 | 50
Nausea (Gastrointestinal disorders) | 99 | 94
Stomatitis (Gastrointestinal disorders) | 46 | 33
Vomiting (Gastrointestinal disorders) | 27 | 26
Asthenia (General disorders) | 47 | 38
Fatigue (General disorders) | 53 | 62
Oedema peripheral (General disorders) | 8 | 18
Pyrexia (General disorders) | 31 | 30
Upper respiratory tract infection (Infections and infestations) | 17 | 8
Infusion related reaction (Injury, poisoning and procedural complications) | 31 | 28
Radiation skin injury (Injury, poisoning and procedural complications) | 33 | 34
Alanine aminotransferase increased (Investigations) | 18 | 30
Aspartate aminotransferase increased (Investigations) | 14 | 25
Ejection fraction decreased (Investigations) | 20 | 9
Neutrophil count decreased (Investigations) | 14 | 13
Decreased appetite (Metabolism and nutrition disorders) | 21 | 20
Arthralgia (Musculoskeletal and connective tissue disorders) | 34 | 40
Bone pain (Musculoskeletal and connective tissue disorders) | 11 | 20
Myalgia (Musculoskeletal and connective tissue disorders) | 27 | 28
Dizziness (Nervous system disorders) | 14 | 8
Headache (Nervous system disorders) | 25 | 21
Peripheral sensory neuropathy (Nervous system disorders) | 14 | 20
Insomnia (Psychiatric disorders) | 16 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 14
Alopecia (Skin and subcutaneous tissue disorders) | 196 | 213
Rash (Skin and subcutaneous tissue disorders) | 18 | 10
Hypertension (Vascular disorders) | 19 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes